CLINICAL TRIAL: NCT05136534
Title: Selective Spinal Anesthesia With Hyperbaric Prilocaine Provides Better Perioperative Pain Control Than Local Anesthesia for Ambulatory Inguinal Hernia Repair Without Affecting Discharging Time: a Randomized Controlled Trial
Brief Title: Spinal Versus Local Anesthesia for Hernia Repair
Acronym: SPINOFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14.16 TS ComEt CBM
Record Dates: First submitted 2021-10-21; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Hernia, Inguinal
Keywords: subarachnoid; anesthesia; prilocaine
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Spinal; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): subarachnoid anesthesia wit hyperbaric prilocaine
  Interventions: Procedure: spinal anesthesia
- group B (Active Comparator): local anesthesia + mild sedation
  Interventions: Procedure: local anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — subarachnoid anesthesia with 2% hyperbaric pilicaine
  Arms: group A
Procedure: local anesthesia — (Mepivacaine 2%) performed by the surgeon before skin incision
  Arms: group B

SUMMARY:
patients underwent inguinal hernia repair; Group A patients received Subarachnoid anesthesia; Group B Patients underwent surgery with local anesthesia (Mepivacaine 2%) performed by the surgeon; Pain assessment was performed using a 0-10 Numerical Rating Scale (NRS). Intraoperative pain was assessed every 10 minutes,

DETAILED DESCRIPTION:
All patients underwent inguinal hernia repair with the Trabucco's technique (15), performed by the same surgical team. Every patient was adequately informed of the procedural sequence of anesthesia and surgery and signed informed consent before being enrolled in the study.

For both groups, patients received mild sedation with Midazolam 0.03 mg/kg i.v.; Paracetamol 1 gr and Ketorolac 30 mg i.v. were given before surgery as multimodal pre-emptive analgesia.

Group A Subarachnoid anesthesia was performed with a 27G Whitacre needle at L2-L3 interspace, with patients on the lateral decubitus corresponding to the side of surgery. The introducer was inserted in the middle point of the space between two spinous processes, with a slightly cranial direction. The spinal needle was passed through the introducer and advanced till the subarachnoid space was reached, as confirmed by cerebrospinal fluid outflow.

Subsequently, 60 mg of Prilocaine 2% were administered in the subarachnoid space, with a low-flow injection technique and the needle bevel turned laterally towards the sloping surgical side. Lateral decubitus was maintained for at least 10 minutes (16).

At 15 minutes from spinal anesthesia execution, and before surgery started, sensory and motor block were assessed by ice-test and numerical 0-3 Bromage Scale, respectively.

Group B Patients underwent surgery with local anesthesia (Mepivacaine 2%) performed by the surgeon before skin incision. Further infiltrations of local anesthetic were ensured in case of pain during the surgery, for a maximum of 400 mg of mepivacaine.

In case of uncontrolled pain, fentanyl 50 mcg i.v. was given for a maximum of two intraoperative administrations. If pain persisted, a deep sedation was performed with propofol continuous i.v. infusion.

Pain assessment was performed using a 0-10 Numerical Rating Scale (NRS). Intraoperative pain was assessed every 10 minutes,

ELIGIBILITY:
Inclusion Criteria: indication for inguinal hernia repair; signed informed consent

-

Exclusion Criteria: neurological disorders; allergy to local anesthetics; liver disease; serious cardiac conduction problems; severe anemia; cardiogenic or hypovolemic shock; congenital or acquired methemoglobinemia; primitive changes in coagulation; patients treated with class III antiarrhythmics (amiodarone); patients who did not suspend anticoagulants/antiplatelet agents; pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Pain assessed by NRS | 13 months
  Pain assessment was performed using a 0-10 Numerical Rating Scale (NRS). Intraoperative pain was assessed every 10 minutes,

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Costa, Principal Investigator — Campus Bio-Medico University
Locations (1):
- CampusBioMedico, Rome, Italy

REFERENCES:
- [Derived] Costa F, Pascarella G, Luffarelli P, Strumia A, Biondo G, Piliego C, Alloni R, Agro FE. Selective spinal anesthesia with hyperbaric prilocaine provides better perioperative pain control than local anesthesia for ambulatory inguinal hernia repair without affecting discharging time: a randomized controlled trial. J Anesth Analg Crit Care. 2022 Jan 31;2(1):6. doi: 10.1186/s44158-022-00034-x. PMID 37386519